CLINICAL TRIAL: NCT01795209
Title: Phase 4 Study of Ranibizumab for the Treatment of Visual Impairment Due to Macular Edema Secondary to Branch Retinal Vein Occlusion in Patients With Initial Fair Visual Acuity
Brief Title: Ranibizumab for Macular Edema Secondary to Branch Retinal Vein Occlusion in Patients With Fair Vision
Acronym: RVOFV
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Samsung Medical Center (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Kyu Hyung Park, Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-1207-162-005; B-1207-162-005 (Other: Seoul National University Bundang Hospital)
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Branch Retinal Vein Occlusion; Macular Edema
Keywords: Branch retinal vein occlusion; Macular edema; Ranibizumab
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranibizumab group (Experimental): Patients will receive three monthly injections of 0.5 mg of Lucentis (0.05 ml), followed by retreatment/rescue laser as needed.
  Interventions: Drug: Ranibizumab; Procedure: Rescue laser
- Standard of care group (Sham Comparator): Patients will receive three monthly sham injections, followed by retreatment/rescue laser as needed.
  Interventions: Device: Sham injection; Procedure: Rescue laser

INTERVENTIONS:
Drug: Ranibizumab — Loading dose: three monthly intravitreal injections of ranibizumab 0.5 mg
  Lucentis stop criteria: V/A ≥20/20 and complete disappearance of macular edema
  Retreatment: visual loss of 5 or more letter compared to previous visit
  Other Names: Lucentis(ranibizumab), 3mg/0.3ml
  Arms: Ranibizumab group
Device: Sham injection — Three monthly sham injections followed by retreatment (sham injections) as needed
  Stop criteria: V/A ≥20/20 and complete disappearance of macular edema
  Retreatment: visual loss of 5 or more letter compared to previous visit
  Arms: Standard of care group
Procedure: Rescue laser — In the Lucentis group: performed if BCVA < 20/40 or CFT ≥ 350um despite of 3 sessions of previous Lucenis injection from Month 6
  In the standard of care group: performed if BCVA < 20/40 or CFT ≥ 350um from Month 3

SUMMARY:
The purpose of this study is to determine the effect of ranibizumab for the treatment of macular edema (ME) secondary to branch retinal vein occlusion (BRVO) in patients with initial fair visual acuity.

DETAILED DESCRIPTION:
Lucentis was approved for ME due to BRVO based on the results from BRAVO study. The inclusion criteria in BRAVO was "best corrected visual acuity (BCVA) 20/40 to 20/320". Therefore, the patients with VA better than 20/40 who are out of inclusion criteria of BRAVO study had no treatment and just wait to reach spontaneous improvement. But, there is unmet needs of these patients and, in actual clinical practice, many retina specialists treat these patients with Ranibizumab. These patients have been experiencing VA improvement after the injection. Based on these clinical backgrounds, the investigator wants to suggest the treatment guidelines in these patients group, which is, early treatment of ranibizumab would be effective and increase patients' QOL. In other words, there are many experiences in these cases among ophthalmologists, but there have been no clinical trials that can endorse the treatments. To confirm the efficacy of ranibizumab in patients with initial fair vision, the investigators started the prospective randomized clinical trial on the efficacy and safety of ranibizumab for the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Foveal center-involving macular edema secondary to BRVO diagnosed within 12 months before study enrollment
2. ETDRS chart BCVA: 63 to 77 letters (20/32 to 20/50 Snellen equivalent)
3. CFT >= 300 um (mean of measurements obtained at screening and Day 0)
4. Signed consent informed
5. male or female, age ≥18 years old

Exclusion Criteria:

1. Prior episode of RVO: Past history of RVO in the study eye diagnosed before 1 year of study enrollment.
2. BCVA improvement >10 letters between screening and Day 0
3. History of other ocular diseases (e.g. diabetic retinopathy, age-related macular degeneration)
4. Laser treatment within 3 months before baseline
5. Intraocular corticosteroid use within 3 months before baseline
6. Anti-vascular endothelial growth factor (VEGF) treatment in the study or fellow eye within 3 months before baseline
7. Intraocular surgery other than cataract surgery, Cataract surgery within 6 months before baseline
8. Stroke or myocardial infarction ≤3 months before baseline
9. Pregnancy or plan to have baby in female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Time to achieve an improvement of 10 or more Early Treatment Diabetic Retinopathy Study (ETDRS) letters in best-corrected visual acuity | 1 year

SECONDARY OUTCOMES:
Mean change from baseline ETDRS letter score over time | 6 months and 1 year
Percentage of patients gaining 10 or more letters in ETDRS letter score from baseline BCVA | 6 months and 1 year
Percentage of patients gaining < 10 letters in ETDRS letter score from baseline BCVA | 6 months and 1 year
Percentage of patients losing < 10 letters in ETDRS letter score from baseline BCVA | 6 months and 1 year
Proportion of patients with who at least maintain baseline BCVA | 6 months and 1 year
Percentage of patients with central foveal thickness (CFT) of < 300 um | 6 months and 1 year
Safety outcomes | 6 months and 1 year
  Frequency, type, and severity of adverse reactions
Mean change from baseline CFT over time | 6 months and 1 year
Mean change from baseline in National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) distance activities subscale score | 6 months and 1 year
Mean change from baseline in contrast sensitivity | 6 months and 1 year
Mean change from baseline in multifocal electroretinogram (mfERG) P1 amplitude | 6 months and 1 year
Percentage of patients losing 10 or more letters in ETDRS letter score from baseline BCVA | 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Hyung Park, M.D., Principal Investigator — Seoul National Univeristy Bundang Hospital; Se Woong Kang, M.D., Principal Investigator — Samsung Medical Center
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam, Gyunggi-do
  - Samsung Medical Center, Seoul

REFERENCES:
- [Background] Campochiaro PA, Heier JS, Feiner L, Gray S, Saroj N, Rundle AC, Murahashi WY, Rubio RG; BRAVO Investigators. Ranibizumab for macular edema following branch retinal vein occlusion: six-month primary end point results of a phase III study. Ophthalmology. 2010 Jun;117(6):1102-1112.e1. doi: 10.1016/j.ophtha.2010.02.021. Epub 2010 Apr 15. PMID 20398941